CLINICAL TRIAL: NCT07237932
Title: Classifications of Adenomyosis and Correlation of Phenotypes in Imaging and Histopathology to Clinical Outcomes
Brief Title: Adenomyosis Imaging,Histo, Clinical
Acronym: adeno I/H/C
Status: Enrolling by invitation | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Samaa Kamal Ahmed Hussien, Resident, Kafrelsheikh University
Other Study IDs: KFSIRH200-573
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to identify and compare the results of imaging studies and evaluating adenomyosis features and post hysterectomy results and their clinical relievants as well as to describe classification for adenomyosis based on one or a combination of clinical, imaging and histopathological features.

Main questions it aim to answer:

What's the relation between clinical symptoms ,maging and histopathological classification of adenomyosis? Research will identify relationships between clinical symptoms, imaging and histopathological classification of adenomyosis Participants will undergo transvaginal ultrasound, non contrast pelvic MRI, hysterectomy then histopathological examination for their uterus

ELIGIBILITY:
Inclusion Criteria:

Age from 35 to 55 years old female Multipara women No previous treatment for uterine adenomyosis within three months Women with heavy menstrual bleeding and dysmenorrhoea Women who completed their families Patient failed medical treatment and hysterectomy is the only remaining line for treatment -

Exclusion Criteria:

Patients not candidate for hysterectomy Positive pregnancy test Patients with contraindications for MRI such as patients with pacemakers, claustrophobia,or other implanted electronic devices Inadequate image quality due to motion artifact

-

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patient multipara complete their family who has heavy menstrual bleeding due to adenomyosis with failure of medical treatment
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Classifications of adenomyosis | 12 months
  Class of adenomyosis according to imaging, histopathology and clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr elsheikh university, Kafr ash Shaykh, Egypt